CLINICAL TRIAL: NCT02707627
Title: A Controlled Trial Investigating the Use of Laser Therapy to Improve Pediatric Burn Scars.
Brief Title: Laser Therapy for Pediatric Burn Scars
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Joel Fish, Medical Director, Burn Program, The Hospital for Sick Children
Other Study IDs: Hospital for Sick Children
Record Dates: First submitted 2016-03-03; First posted 2016-03-14 (Estimated); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Cicatrix, Hypertrophic; Burns
Keywords: Pediatric; Laser; Burn; Scar; Photothermolysis
MeSH Terms: conditions — Cicatrix, Hypertrophic; Burns; Cicatrix | interventions — Laser Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Laser Therapy: Participants will receive laser therapy for the treatment of their hypertrophic burn scars. Laser treatment decisions will be tailored to meet the needs of the patient.
  Interventions: Device: Laser Therapy

INTERVENTIONS:
Device: Laser Therapy — Laser therapy is a technology that can be used to treat hypertrophic burn scars.

SUMMARY:
A new era of outcomes for pediatric burn patients has begun as burn care continues to improve. Unfortunately, complete restoration of burn-injured skin may be limited by the development of hypertrophic scarring. Treatment with laser therapy is one of the newest forms of scar therapy available. Although laser therapy has only been adopted by burn clinicians within the last several years, early evidence suggests that it may offer significant benefits. Thus the aim of this study is to investigate the effectiveness of using laser therapy to treat hypertrophic burn scars in pediatric patients by using a comprehensive set of subjective and objective scar assessment tools.

ELIGIBILITY:
Inclusion Criteria:

1. Age 1-18 years at presentation
2. Patients with a hypertrophic burn scar that has been clinically diagnosed by a burn care specialist
3. Hypertrophic burn scar resulting from any etiology
4. Hypertrophic burn scar is ≥ 2 months post healing
5. Ability to complete English- language questionnaires

Exclusion Criteria:

1. Patients with concomitant skin disease (i.e. chronic skin conditions, herpes infection)
2. Patients with a history of keloid scarring
3. Patients who cannot tolerate the intravenous (IV) sedation used to perform laser therapy procedures
4. Patients who have had previous laser therapy procedures

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Eligible participants will be pediatric patients with hypertrophic scars requiring treatment.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-10; Primary Completion 2020-05 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Vancouver Scar Scale Score | Baseline (month 0) to month 12
  The Vancouver Scar Scale is composed of four subscales which include pigmentation (range: 0 - 3), vascularity (range: 0 - 3), pliability (range: 0 - 5), and height (range: 0 - 3).
  Total Vancouver Scar Scale score refers to the score obtained by summing the values from each subscale (range: 0 - 14) with higher scores indicating a worse scar.

SECONDARY OUTCOMES:
Patient and Observer Scar Assessment Scale Score | Baseline (month 0) to month 12
  The Patient and Observer Scar Assessment Scale consists of two independent scales: 1) the patient scale (patient-reported), and 2) the observer scale (clinician-reported). Both the patient scale as well as the observer scale include a set of individual subscales that assess scar severity (range: 1 - 10) with higher scores indicating a worse scar.
Scar thickness | Baseline(month 0) to month 12
  Scar thickness measurements will be taken at five study visits over the course of one year and will be measured using ultrasonography.
Scar stiffness measured by the DermaLab Combo® skin analysis device | Baseline(month 0) to month 12
  Scar stiffness measurements will be taken at five study visits over the course of one year and will be measured using the DermaLab Combo® skin analysis device (Cortex Technologies, Hadsund, DK).
Scar stiffness measured by ultrasound elastographgy | Baseline(month 0) to month 12
  Scar stiffness measurements will be taken at five study visits over the course of one year and will be measured using ultrasound elastography.
Scar colour | Baseline(month 0) to month 12
  Scar colour measurements will be taken at five study visits over the course of one year and will be measured using the DermaLab Combo® skin analysis device (Cortex Technologies, Hadsund, DK)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada